CLINICAL TRIAL: NCT01839968
Title: Ex-Vivo Reversion of Platelet Inhibition Induced by Prasugrel
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Fanny Bonhomme, MD, University Hospital, Geneva
Other Study IDs: 11-117
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Acquired Platelet Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma

GROUPS / COHORTS (1):
- Study patients: Acute coronary syndrome patients with a recent loading dose of prasugrel (6-24h)
  Interventions: Other: Ex vivo addition of normal platelet rich plasma to prasugrel-treated platelet rich plasma

INTERVENTIONS:
Other: Ex vivo addition of normal platelet rich plasma to prasugrel-treated platelet rich plasma

SUMMARY:
The purpose of this ex-vivo study is to estimate the optimal platelet quantity necessary to reverse the antiplatelet effects of prasugrel.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome
* Prasugrel loading dose 6-24h before inclusion

Exclusion Criteria:

* Clopidogrel loading dose
* GPIIbIIIa use within 10 days before inclusion
* Known congenital thrombopathy and/or congenital coagulation defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome who received a loading dose of prasugrel within 6 and 24h.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity assessed by light transmittance aggregometry (LTA) after ex-vivo normal platelet addition | within the first 6-24 hours after antiplatelet drug loading dose

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland